CLINICAL TRIAL: NCT03460613
Title: Prevalence of FODMAP Intolerance and Joint Hypermobility Syndrome in Functional Bowel Patients and Association With Microbiome, Dyssynergic Defecation and Dietary Intervention - a Prospective Cohort Study With Health-related Intervention
Brief Title: Prevalence of FODMAP Intolerance and JHS in FGID and Association With Microbiome, Dyssynergic Defecation and Dietary Intervention
Acronym: PreDiMi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-01887
Record Dates: First submitted 2017-07-06; First posted 2018-03-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FGID Patients (Other)
  Interventions: Other: FODMAP diet
- Hepatology Control Group (No Intervention)
- Healthy Volunteers (No Intervention)

INTERVENTIONS:
Other: FODMAP diet — Patients with a diagnosed FODMAP intolerance (and a control with no FODMAP intolerance) by prior nutrient challenge testing are going on a FODMAP diet or a 2-food elimination diet (wheat products, milk products excluded).
  For the FODMAP diet: In a first nutritional visit a specialized nutritionist will inform the patients about FODMAP containing foods and illustrate a FODMAP elimination diet. After 3 weeks of elimination diet another visit will take place and a stepwise reintroduction diet is initiated after successful elimination diet. For the 2-food elemination diet: In a first nutritional visit a specialized nutritionist will inform the patients about the 2-food-elimination diet (foods containing milk- and wheat products) and illustrate an elimination diet. After 3 weeks of elimination diet another visit will take place and a stepwise reintroduction diet is initiated after successful elimination diet.
  Arms: FGID Patients

SUMMARY:
Irritable bowel syndrome (IBS) is a disorder of gastrointestinal function characterized by abdominal symptoms and pain associated with alterations in bowel habit. The condition impacts on the quality of life of at least 10% of the population, impacts on activities of daily living and is associated with considerable direct and indirect costs to the individual, the health system and society. The etiology of IBS appears multifactorial and several mechanisms, among them mucosal inflammation, abnormal intestinal motility, visceral hypersensitivity and psychological factors, appear to be involved.

An underlying pathophysiology, namely Joint Hypermobility (JH) and Joint Hypermobility Syndrome (JHS), that we are going to study, have recently gained increasing attention in patients with functional bowel disease.

One factor which was shown in previous IBS-studies to reduce abdominal symptoms is a FODMAP diet.

To identify FGID patients which profit most from different diagnostics and therapies (such as dietary intervention (FODMAP diet, 2-food-elimination diet)) we are going to carry out a study analyzing different subtypes of FGID (in particular IBS, FD, functional abdominal pain/bloating) for demographics, clinical diagnostics (e.g. nutrient challenge testing, microbiome testing, anorectal manometry and MR defecography), comorbidities (in particular JH, JHS and psychological comorbidities) and treatment.

DETAILED DESCRIPTION:
Functional gastrointestinal disorders (FGID) are common in the general population. Symptoms such as pain, nausea, bloating, diarrhea or constipation may occur. Irritable bowel syndrome (IBS) is the most common FGID with a prevalence in the range of 5-25%. Medical attention is sought by 20-75% of patients who meet diagnostic criteria for IBS at some time in their lives. Quality of life is often impaired in IBS patients. In previous studies a diet low in FODMAP was shown to reduce gastrointestinal symptoms in IBS patients.

But still it is unknown which FGID patients (e.g. patients with irritable bowel syndrome, functional dyspepsia (FD), functional abdominal pain/bloating) profit most from such a diet which involves costs, time and significant lifestyle alteration.

To test for food intolerances, standard hydrogen breath tests using fructose or lactose as challenge substance are still commonly used and do present a nutritional challenge, however the usefulness of information gained is questionable. Fructose intolerance is as prevalent in IBS as in healthy volunteers, in fact when tested with the usual doses of 25-50g, prevalence of fructose intolerance ranges between 53% and 73%. Testing (genetic) for hypolactasia, is often, even in the professional setting, misunderstood as lactose intolerance testing. Most patients, who do have hypolactasia, i.e. almost no activity of intestinal brush-border enzyme lactase, tolerate up to 12g of lactose per day, remain asymptomatic and therefore should not be considered lactose intolerant. In addition, one must realize, that the vast majority in the world is hypolactasic and hypolactasia, or rather lactase persistence, constitutes a norm variant.

Recently it was shown that a standardized liquid mixed nutrient meal including 25g lactulose, but not with 15g lactulose, allows differentiation of IBS patients from healthy controls. This test, incorporating FODMAP lactulose, that, unlike lactose and fructose, is indigestible in all humans in the small intestine, plus a caloric load, reflecting a regular meal and everyday life, has therefore the potential to be a useful marker of nutrient intolerance in patients with suspected functional bowel disease.

Additionally, associations between FGID and JH/JHS have been recognized in the past decade. JH/JHS constitutes a hereditary disorder of connective tissue in which patients often report non-musculoskeletal symptoms, among them gastrointestinal complaints. Previous studies in Europe and the U.S. have reported a JHS prevalence of 20% in the general population.

A stringent approach to studying possibly JH and JHS-related changes with diagnostic and interventional arms, such as a nutrient challenge testing or dietary adaptation (i.e.FODMAP diet, 2-food-elimination diet) has not yet been taken.

Differences in the intestinal microbiome have been shown in IBS patients compared to healthy volunteers but not in JHS compared to non-JHS patients. Given the differences noted in patients' symptomatology, the preliminary data on gut function and the underlying structural abnormalities, the role of microbiome in relation to FGID and JHS is highly interesting and, as yet, unstudied. In recent years with the advent of more powerful sequencing tools, a number of studies have been published, that try to characterize the microbiome in IBS patients. Research on IBS-related changes of the microbiome is early and incomplete. The number of literature reviews regarding gut microbiome currently far exceeds the number of original articles reporting on the microbiome in functional bowel disease. IBS-specific interventional studies are even rarer and when performed, often lack control groups and the reality of multiple or repeated intervention, that characterize treatment of FGID. Therefore, and to identify patients according to their microbiome which profit most from therapeutic intervention (such as FODMAP diet, 2-food elimination diet) we are also going to analyze microbiome changes before and after dietary intervention.

Another pathological, impairing aspect of IBS patients is the intestinal hypersensitivity. Anorectal hypersensitivity measurement has been considered a hallmark for IBS for many years. We are routinely performing anorectal functions tests in our specialized unit. Recently we validated high-resolution anorectal manometry and rapid barostat bag measurements to assess visceral sensitivity; in a further study we assessed obstructive defecation when compared to magnetic resonance defecography. In an earlier study employing magnetic resonance defecography (MR defecography) we were able to show that MR defecography, apart from correlating well with the diagnosis of dyssynergic defecation suggested by anorectal manometry, additional pelvic floor abnormalities such as pelvic floor descent, cystocele and enterocele could be identified. Studying these measures in patients with suspected outlet obstruction in relation to JHS status, which is considered a risk factor for pelvic floor abnormalities, might lead to more focused diagnostic and therapeutic approaches in the future for patients who profit most from certain procedures.

Considering all above mentioned facts we are going to carry out a study analyzing different subtypes of FGID (in particular IBS, FD, functional abdominal pain/bloating) for demographics, clinical diagnostics (e.g. nutrient challenge testing, microbiome testing, anorectal manometry and MR defecography), treatment (FODMAP diet) and comorbidities (in particular JH, JHS and psychological comorbidities) to identify FGID patients which profit most from different diagnostics and dietary interventions.

ELIGIBILITY:
Inclusion criteria for FGID patients:

* Functional bowel disease as per physician's diagnosis (medical judgement) and Rome IV criteria
* Signed Informed Consent after being informed
* Age 18-60 years

Inclusion criteria for hepatology control cohort:

* Signed Informed Consent after being informed
* Age 18-60 years
* Patient in the ambulatory hepatology clinic

Inclusion criteria for healthy volunteers:

* Signed informed consent after being informed
* Age 18-60 years

Exclusion criteria for FGID patients:

* Inflammatory bowel disease
* Gastrointestinal malignancy
* Celiac Disease
* Known or suspected non-compliance, drug or alcohol abuse
* Previous large abdominal surgery likely to impact patient symptomatology
* Inability to follow the procedures of the study, e.g. due to language problems, dementia, etc. of the participant
* Previous enrollment into the current study
* Use of antibiotics in the previous 4 weeks before enrolment

Exclusion criteria for hepatology control cohort:

* Previous diagnosed functional gastrointestinal disorders

Exclusion criteria for healthy volunteers:

* Previous diagnosed functional gastrointestinal disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 498 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of Joint Hypermobility / hypermobile Ehlers-Danlos Syndrome according to the criteria of the "2017 International Classification of the Ehlers-Danlos Syndromes" (hEDS) | 15 minutes
  Prevalence of joint hypermobility resp. hEDS will be assessed by physicians according to the criteria of the "2017 International Classification of the Ehlers-Danlos Syndromes" in patients with disorders of gut-brain interactions (FGID). The assessment consists of some hypermobility testings (wrists, fingers, elbows, knees and legs) and questions about family hypermobility syndrome history, scars healing, hernia history etc.

SECONDARY OUTCOMES:
Prevalence of FODMAP intolerance according to nutrient challenge testing (NCT). | 3-4 hours
  Prevalence of FODMAP intolerance in FGID patients will be assessed according to nutrient challenge testing (NCT). Patients drink a specific beverage containing a specific sugar. The hydrogen value in breath is then measured every 10 minutes and symptoms are recorded at the same time. Depending on the time of hydrogen production and the increase of abdominal symptoms can a FODMAP intolerance be determined.
Response to dietary intervention | 10-12 weeks
  FGID patients will be randomized according to the participants JH-status and according to the result of NCT to the dietary intervention. Patients will be randomised to a low FODMAP-diet or 2-food-elimination diet. They will follow a specific intervention diet with guidance of a dietician and the abdominal symptoms will be assessed every 4 weeks approximately.

OTHER OUTCOMES:
Microbiome in FGID patients | 3-4 weeks
  Microbiome changes after dietary intervention will be analyzed.
Prevalence of outlet obstruction in IBS-C subgroup | 1-3 hours
  Prevalence of outlet obstruction in a subgroup of FGID patients (IBS-C) will be analyzed by high resolution anorectal manometry and/or MR defecography

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pohl, PD Dr. med., Principal Investigator — University of Zurich
Locations (1):
- UniversitätsSpital, Zurich, Switzerland